CLINICAL TRIAL: NCT00885508
Title: A Phase II Study of the Efficacy and Safety of Lenalidomide Combined to Escalating Doses of Chemotherapy in Intermediate-2-or High Risk MDS and AML With Del 5q
Brief Title: A Study of the Efficacy and Safety of Lenalidomide Combined to Escalating Doses of Chemotherapy in Intermediate-2-or High Risk Myelodysplastic Syndrome (MDS) and Acute Myeloid Leukemia (AML) With Del 5q
Acronym: GFM-Chimio-Rev
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GFM-Chimio-Rev-08; NCT00922298 (obsolete NCT alias)
Record Dates: First submitted 2009-04-21; First posted 2009-04-22 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Myelodysplastic Syndrome; Chronic Myelomonocytic Leukemia; Acute Myeloid Leukemia
Keywords: MDS; AML; deletion 5q; Documented diagnosis of MDS, or CMML; with WBC < 13,000/mm3 that meets IPSS criteria for intermediate-2; or high-risk disease, or AML with an associated del 5q[31]; (the deleted chromosomal region must include 5q[31]),; with or without additional cytogenetic abnormalities
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Acute | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aracytidine, Daunaurubicine, Lenalidomide (Experimental)
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — 1. Induction treatment Lenalidomide 10 mg once daily PO during 3 weeks . in combination with classical 7+3 chemotherapy.
  2. Consolidation treatment 6 monthly courses of : Lenalidomide 10 mg/ d during the first 2 weeks in combination with classical 5+1 consolidation chemotherapy
  3. Maintenance treatment Lenalidomide 10 mg/d 2 weeks every month until relapse
  In absence of toxicity, 20 additionnal patients will be included with lenalidomide dose of 25mg/J, then 20 other additionnals patients with Lenalidomide 50mg/J

SUMMARY:
In this trial, the investigators will test the combination of escalating doses of chemotherapy (starting at relatively low dose) with lenalidomide in intermediate-2-or high risk MDS and AML with del 5 q31. It is hoped that this combined therapy will further increase response rate in intermediate-2-or high risk MDS and AML with del 5 q31, without major toxicity in comparison to historical results obtained with chemotherapy alone in the same subset of patients.

DETAILED DESCRIPTION:
Patients will receive lenalidomide combined to DNR- AraC chemotherapy. The first 31 patients will receive DNR 45 mg/m2/d, during 3 days, and AraC 200mg/m2/d CI during 7 days.

Progression or not to the next cohort DNR 60 mgm2/d x3d and AraC 200mg/m2d x7d , or on the contrary reduction to the lower cohort DNR 30 mgm2/d x3d and AraC 200mg/m2d x5d will be decided after inclusion of fixed numbers of patients ,after review of toxicity and efficacy by an independent safety review committee (SRC).

Efficacy would be defined as a response rate ≥50%. After inclusion of the first 31 patients, the SRC will choose the cohort dose the last 33 patients will receive, based on toxicity and efficacy criteria.

1. Induction treatment Lenalidomide 10 mg once daily PO during 3 weeks . DNR 30-45-or 60 mg/m2 /d (depending on the cohort during 3 days (IV push)- AraC 200mg/m2/d during 5- 7 or 7 days (continuous infusion)+ G-CSF (lenograstim): 263 ug/d from day 9, until recovery from aplasia (maximum 30 days).

   Evaluation will be performed after recovery from aplasia, on day 40 at the latest (with marrow aspirate and karyotype).

   Patients in hematological CR, CRi or marrow CR will proceed to consolidation treatment

   :Once the cohort dose has been decided by the SRC, a second cohort of 33 patients will be enrolled
2. Consolidation treatment (in patients who achieved CR, Cri, or marrow CR) 6 monthly courses of : DNR (at the daily dose required to achieve CR) day1, combined to AraC 60 mg/m2/12h SC during 5 days will be given.

   Lenalidomide 10 mg/ d during the first 2 weeks of the course.
3. Maintenance treatment Lenalidomide 10 mg/d 2 weeks every month until relapse (dose reduced if cytopenias) In patients still responding after 52 weeks, the drug will continue to be supplied, and follow up until death will be continued in all patients.

SECOND PART OF THE TRIAL AFTER AMENDMENT Treatment schedule of the 2nd Part of the trial

In dose level 4, 20 patients will receive lenalidomide 25 mg/d during 21 days combined to DNR- AraC chemotherapy (DNR 60 mgm2/d x3d and AraC 200mg/m2d x7d) during induction. During consolidation, patients will receive Lenalidomide 25 mg/d during 14 days, combined with DNR 60 mgm2/d x1d and AraC 60 mg/m2 x2/d x5d. finally, during maintenance, patients will receive Lenaidomide 25 mg/d x14d every months, until relapse.

Progression or not to the next cohort (Lenaidomide 50 mg) will be decided after inclusion of 20 patients, after review of toxicity and efficacy by an independent safety review committee (SRC) (Briefly, given median times to reach ANC and platelets > 500 and 50000/mm3, respectively of about 27 days in our previous trial with chemotherapy alone (Gardin, Blood), DLT would be defined by having greater than 3 of 10 patients recovering those levels after more than 40 days, or the occurrence of unexpected grade III-IV non hematological toxicity). Efficacy would be defined as a response rate ≥60%.

In dose level 5, 20 patients will receive lenalidomide 50 mg/d during 21 days combined to DNR- AraC chemotherapy (DNR 60 mgm2/d x3d and AraC 200mg/m2d x7d) during induction. During consolidation, patients will receive Lenalidomide 50 mg/d during 14 days, combined with DNR 60 mgm2/d x1d and AraC 60 mg/m2 x2/d x5d. finally, during maintenance, patients will receive Lenaidomide 50 mg/d x14d every months, until relapse.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Must understand and voluntarily sign an informed consent form
3. Must be able to adhere to the study visit schedule and other protocol requirements
4. No contra indication to anthracycline based chemotherapy
5. Documented diagnosis of MDS, or CMML with WBC < 13,000/mm3 that meets IPSS criteria for intermediate-2 or high-risk disease, or AML with an associated del 5q[31] (the deleted chromosomal region must include 5q[31]), with or without additional cytogenetic abnormalities
6. Female subjects of childbearing potential must:

   * Understand that the study medication could have a potential teratogenic risk
   * Agree to use, and be able to comply with, effective contraception without interruption, 4 weeks before starting study drug, throughout study drug therapy (including dose interruptions) and for 4 weeks after the end of study drug therapy, even if she has amenorrhoea. This applies unless the subject commits to absolute and continued abstinence confirmed on a monthly basis. The following are effective methods of contraception:

     * Implant, Levonorgestrel-releasing intrauterine system (IUS) (prophylactic antibiotics should be considered at the time of insertion particularly in patients with neutropenia due to risk of infection) , Medroxyprogesterone acetate depot, Tubal sterilization, Ovulation inhibitory progesterone-only pills (i.e., desogestrel), Sexual intercourse with a vasectomised male partner only; vasectomy must be confirmed by two negative semen analyses.
     * Combined oral contraceptive pills are not recommended. If a subject was using combined oral contraception, she must switch to one of the methods above. The increased risk of VTE continues for 4 to 6 weeks after stopping combined oral contraception.
   * Agree to have a medically supervised pregnancy test with a minimum sensitivity of 25 mIU/ml not more than 3 days from the start of study medication once the subject has been on effective contraception for at least 4 weeks. This requirement also applies to women of childbearing potential who practice complete and continued abstinence.
   * Agree to have a medically supervised pregnancy test every 4 weeks including 4 weeks after the end of study treatment, except in the case of confirmed tubal sterilization. These tests should be performed not more than 3 days before the start of next treatment. This requirement also applies to women of childbearing potential who practice complete and continued abstinence
7. Male subjects must:

   * Agree to use condoms throughout study drug therapy, during any dose interruption and for one week after cessation of study therapy if their partner is of childbearing potential and has no contraception.
   * Agree not to donate semen during study drug therapy and for one week after end of study drug therapy.
8. All subjects must:

   * Agree to abstain from donating blood while taking study drug therapy and for one week following discontinuation of study drug therapy.
   * Agree not to share study medication with another person and to return all unused study drug to the investigator

Exclusion Criteria:

1. Pregnant or lactating females.
2. Contra indication to anthracycline based chemotherapy.
3. Proliferative (WBC ≥ 13,000/mL) CMML.
4. Prior ≥ grade-2 NCI CTCAE (v 3.0) allergic reaction to thalidomide.
5. Prior desquamating (blistering) rash while taking thalidomide.
6. Prior history of malignancy other than MDS unless the subject has been free of disease for ≥ 5 years.
7. Use of cytotoxic chemotherapeutic agents or experimental agents (agents that are not commercially available) for the treatment of MDS within 28 days .
8. Less than 6 months since prior allogeneic bone marrow transplantation.
9. Less than 3 months since prior autologous bone marrow or stem cell transplantation.
10. Recombinant human erythropoietin (rHuEPO) therapy received within 28 days.
11. Known HIV-1 positivity.
12. Any serious medical condition or psychiatric illness that will prevent the subject from signing the informed consent form or will place the subject at unacceptable risk if he or she participates in the study.
13. Creatinine Clearance< 50 ml/min
14. Serum aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) or alanine transaminase (ALT)/serum glutamate pyruvate transaminase (SGPT) > 3.0 x upper limit of normal (ULN)
15. Serum total bilirubin > 1.5 mg/dL (expect for unconjugated hyperbilirubinemia due to Gilbert's disease or secondary to MDS).
16. Subjects with ≥ grade-2 neuropathy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2009-02; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Response (CR, mCR and Cri, according to IWG criteria for AML and IWG 2006 criteria for MDS) to the combination of lenalidomide and chemotherapy in adult high and int 2 MDS (IPSS) or AML with deletion 5q[31] | At the end of induction

SECONDARY OUTCOMES:
Duration of response | At 1 and 2 years
Progression to AML | At 1 and 2 years
Survival and safety of the combination of lenalidomide and chemotherapy | At 1 and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lionel Adès, MD, Principal Investigator — Groupe Francophone des Myelodysplasies
Locations (25):
- France (25):
  - CH Angers, Angers
  - hopital Victor Dupouy, Argenteuil
  - Centre Hospitalier de La Cote Basque, Bayonne
  - Hôpital Avicenne, Bobigny
  - CHU Haut-Lévèque, Bordeaux
  - Centre hospitalier de Chambéry, Chambéry
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - Centre henri Mondor, Créteil
  - Centre Hospitalier du Mans, Le Mans
  - Centre Hospitalier de Lens, Lens
  - centre hospitalier de Lens, Lens
  - Hôpital Limoges, Limoges
  - Centre Hospitalier Lyon Sud, Lyon
  - Institut Paoli Calmettes, Marseille
  - CHU Brabois, Nancy
  - CHU de nantes, Nantes
  - Hôpital Archet1, Nice
  - Hoiptal St Louis, Paris
  - Hopital Cochin-Hematology, Paris
  - Centre Hospitalier Joffre, Perpignan
  - Centre Henri Becquerel, Rouen
  - Hôpital Hautepierre, Strasbourg
  - Hopital Purpan Service d'Hématologie Clinique, Toulouse
  - CH de Valence, Valence
  - Institut gustave Roussy, Villejuif

REFERENCES:
- [Derived] Ades L, Prebet T, Stamatoullas A, Recher C, Guieze R, Raffoux E, Bouabdallah K, Hunault M, Wattel E, Stalnikiewicz L, Toma A, Dombret H, Vey N, Sebert M, Gardin C, Chaffaut C, Chevret S, Fenaux P. Lenalidomide combined with intensive chemotherapy in acute myeloid leukemia and higher-risk myelodysplastic syndrome with 5q deletion. Results of a phase II study by the Groupe Francophone Des Myelodysplasies. Haematologica. 2017 Apr;102(4):728-735. doi: 10.3324/haematol.2016.151894. Epub 2016 Dec 29. PMID 28034993
- See also: Website of the french group of MDS — http://www.gfmgroup.org